CLINICAL TRIAL: NCT02852525
Title: Real-Time Evaluation of Barrett's Esophagus by Confocal Laser Probe-based Microscopy
Brief Title: Confocal Laser Probe to Treat Barrett's Esophagus
Acronym: pCLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virendra Joshi (Other)
Responsible Party: Sponsor-Investigator, Virendra Joshi, Virendra Joshi,MD, Ochsner Health System
Organization: Ochsner Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Barrett's Confocal
Record Dates: First submitted 2014-01-21; First posted 2016-08-02 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-07

CONDITIONS: Barrett's Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Confocal laser endomicroscopy (pCLE) (Other): Patients agreeing to participate in the research study will receive an additional intravenous injection during endoscopy. This dose of 2.5 mg of IV fluorescein will be administered during their EGD. Probe-based microscopy will be used to evaluate the mucosa of the esophagus and GE junction. Photographs will be taken and digitally stored. Biopsies (which are part of the routine diagnosis and surveillance of Barrett's) will be targeted based on the microscopic images. The histologic findings on the biopsy specimens will be compared to the microscopic images to determine the accuracy of the probe-based microscopy in predicting pathology.
  Interventions: Device: Confocal laser endomicroscopy (pCLE)

INTERVENTIONS:
Device: Confocal laser endomicroscopy (pCLE) — Patients agreeing to participate in the research study will receive an additional intravenous injection during endoscopy. This dose of 2.5 mg of IV fluorescein will be administered during their EGD. Probe-based microscopy will be used to evaluate the mucosa of the esophagus and GE junction

SUMMARY:
The purpose of this study is to further validate the use of probe-based confocal laser endomicroscopy (pCLE) for the evaluation of Barrett's Esophagus and associated neoplasia in a larger patient base.

DETAILED DESCRIPTION:
Subject Population

Approximately 100 subjects will be recruited, age greater than 18 years. Subjects will be recruited from OCF, OMC Kenner who are undergoing EGD for either 1) screening for Barrett's Esophagus because of long-standing GERD of greater than 5 years; 2) surveillance of known Barrett's Esophagus; or 3) therapy for known Barrett's Esophagus. They will be asked to volunteer for participation at the time of their EGD. These subjects are being recruited because of a high suspicion or known diagnosis of Barrett's Esophagus in this cohort.

Procedures

Patients agreeing to participate in the research study will receive an additional intravenous injection during endoscopy. This dose of 2.5 mg of IV fluorescein will be administered during their EGD. Probe-based microscopy will be used to evaluate the mucosa of the esophagus and GE junction. Photographs will be taken and digitally stored. Biopsies (which are part of the routine diagnosis and surveillance of Barrett's) will be targeted based on the microscopic images. The histologic findings on the biopsy specimens will be compared to the microscopic images to determine the accuracy of the probe-based microscopy in predicting pathology.

The time commitment for the patient is included in the time to undergo endoscopy and is roughly 30 minutes to an hour, including recovery time. The research will occur at OMC, Jefferson Highway and Ochsner Medical Center, Kenner.

ELIGIBILITY:
Inclusion Criteria:

* Must be greater than 18 years of age
* currently undergoing EGD
* previous diagnosis of Barrett's Esophagus
* long-standing GERD of greater than 5 years
* undergoing therapy for previously diagnosed Barrett's Esophagus

Exclusion Criteria:

* Under 19 years of age

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of probe based endomicroscopy as compared to histopathology in diagnosing Barrett's metaplasia | 30 minutes up to an hour on average after undergoing endoscopy

SECONDARY OUTCOMES:
Tissue and blood Biomarker evaluation in targeted biopsies obtained at endomicroscopy in patients diagnosed to have Barrett's metaplasia and dysplasia | 30 minutes up to an hour on average after undergoing endoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Virendra Joshi, MD, Principal Investigator — Ochsner Health System
Locations (2):
- United States (2):
  - Oschsner Medical Center-Kenner, Kenner, Louisiana
  - Ochsner Medical Center-Jefferson Highway, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: Undecided